CLINICAL TRIAL: NCT04333732
Title: An International, Multi-site, Bayesian Platform Adaptive, Randomized, Placebo-controlled Trial Assessing the Effectiveness of Candidate Agents in Mitigating COVID-19 Disease in Adults
Brief Title: CROWN CORONATION: COVID-19 Research Outcomes Worldwide Network for CORONAvirus prevenTION
Acronym: CROWN CORONA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: COVID -19 Therapeutics Accelerator (Unknown)
Responsible Party: Principal Investigator, Michael Avidan, Professor of Anesthesiology and Surgery, Washington University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 202004099; INV-017499 (Other Grant/Funding Number: Bill and Melinda Gates Foundation)
Record Dates: First submitted 2020-03-31; First posted 2020-04-03 (Actual); Results first posted 2024-03-26 (Actual); Last update posted 2024-03-26 (Actual); Status verified 2024-01

CONDITIONS: COVID 19
Keywords: COVID 19; Health care workers; M-M-R II ®
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: An international, multi-site, randomized, placebo-controlled, Bayesian platform clinical trial. Initially there will be 2 arms, but we anticipate adding intervention arms to the platform. Combining interventions, allowing assessment of potential interactions, will be considered when arms are added.
Who Masked: Participant, Investigator
Masking Description: For the MR or MMR vaccine, there will be a placebo vaccine. Attempts will be made to maintain masking for other interventions (e.g. oral tablets) added to the platform by including suitable placebo options.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- M-M-R II ® (Experimental): Education and surveillance plus M-M-R II ® Single dose, 0.5 mL subcutaneous injection of M-M-R II ®
  Interventions: Drug: MR or M-M-R II ® vaccine
- Placebo (Placebo Comparator): Education and surveillance plus placebo Single dose, 0.5 mL subcutaneous injection of 0.9% saline
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: MR or M-M-R II ® vaccine — Education and surveillance plus MR or M-M-R II ® vaccine
  Other Names: Merck
  Arms: M-M-R II ®
Drug: Placebo — Placebo injection
  Arms: Placebo

SUMMARY:
The objective of CROWN CORONATION is the prevention of symptomatic COVID-19 by using combinations of approved and safe repurposed interventions, with complementary mechanisms of action.

DETAILED DESCRIPTION:
CROWN CORONATION is an international, Bayesian platform adaptive, randomized, placebo-controlled trial assessing the effectiveness of candidate interventions in preventing COVID-19 disease in adults.

Randomization will be stratified by age (<50 and ≥50) and site. Participants will be healthcare workers at risk of contracting SARS-CoV-2. Participants will be randomized into one of two arms:

* Education and surveillance plus MR or MMR vaccine
* Education and surveillance plus Placebo

While the initial intervention to be tested on the platform will be the MR or MMR vaccine, other interventions might be added or removed over the course of the trial. The trial will evaluate which of the intervention arms is most effective at decreasing the incidence of symptomatic COVID-19 disease, without unacceptable side effects or safety events.

All participants will require be required to have a mobile phone to participate. This is standard in all the countries in this study. Most, but not all, will also have a smartphone. Participants will complete weekly data logs via SMS texting. Follow-up information will be collected until approximately 5 months after the end of treatment or death. Participants who develop symptomatic COVID-19 during the last month of observation will at a minimum be followed-up until symptom resolution and at a maximum until 6 months after randomization (whichever comes first). Telemedicine approaches to collecting information on participants will be used where possible. The trial will provide adherence support interventions that have been shown in randomized controlled trials to improve adherence to Human Immunodeficiency Virus treatment and adapted for HIV Pre-Exposure Prophylaxis (HIV PrEP) (e.g. two-way SMS with check in for those that report symptoms or adverse events). The database will be hosted on UK-based servers which are expected to be managed by Sealed Envelope Ltd. Local investigators will have access to the part of the CRF to enable recording of outcome data and/or severity of COVID-19 symptoms. Participants will be given a secure login to enable them to complete an initial participant health questionnaire and the regular data logs. It is envisaged that these will be completed at least weekly.

ELIGIBILITY:
Inclusion criteria

1. Volunteers without clinical evidence of COVID-19 infection aged 18 years and older.
2. Healthcare workers based in a primary, secondary or tertiary healthcare setting with a high risk of developing COVID-19 due to their potential exposure to patients with SARS-CoV-2 infection.
3. Must have a mobile phone and access to the Internet for data collection purposes.
4. Participants who are willing and able to provide informed consent via an electronic consent process.

Exclusion criteria

1. Prior enrollment into other COVID-19 interventional prevention or treatment trials (observational trials not excluded).
2. Self-reported or diagnosed current infection with SARS-CoV-2 or previous COVID-19 diagnosis.
3. Self-reported current acute respiratory infection.
4. Concurrent and/or recent involvement in other research or use of the investigational product, a product considered to be equivalent to the investigational product, or any other product that is likely to interfere with the investigational products in this trial used within three months of study enrolment.
5. Self-reported known allergies to any of the IMPs and excipients of the IMPs and placebo.
6. Self-reported presence or history of the conditions listed in the appendices.
7. Self-reported current use of medication known to interact with any of the medications listed in the appendices.
8. Inability or unwillingness to be followed up for the trial period.

For M-M-R II

* Pregnant women.
* Individuals receiving high dose corticosteroids, other immuno-suppressive drugs, alkylating agents or anti-metabolites.
* Individuals undergoing radiotherapy.
* Any malignant disease either untreated or currently undergoing therapy.
* History of administration of gammaglobulin or blood transfusions within the previous 3 months.
* Participants with an allergy to the MR (MMR) vaccine or its components, including neomycin.
* Idiopathic thrombocytopenic purpura (ITP)
* Untreated tuberculosis
* Prior receipt of any vaccines (licensed or investigational) ≤30 days before enrollment
* Planned receipt of any vaccine other than the study intervention within 30 days before and after the study vaccination (not including the flu vaccination via injection)
* Prior receipt of an investigational or licensed vaccine likely to impact on interpretation of the trial data (e.g. Adenovirus vectored vaccines, any coronavirus vaccines).
* Any confirmed or suspected immunosuppressive or immunodeficient state, including untreated HIV infection with a CD4T count <200 /mL
* Asplenia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3411 (Actual)
Dates: Start 2020-09-04 (Actual); Primary Completion 2021-08-10 (Actual); Study Completion 2021-12-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael S. Avidan, MBBCh, Principal Investigator — Washington Univeristy School of Medicine; Ramani Moonesinghe, MD, Principal Investigator — University College, London; Helen Rees, MD, Principal Investigator — Wits University
Locations (17):
- Washington University School of Medicine, St Louis, Missouri, United States
- University of Ghana Medical Centre, Accra, Greater Accra Region, Ghana
- South Africa (12):
  - Groote Schuur/J52, Desmond Tutu Health Foundation, Mowbray, Cape Town
  - Masiphumelele, Desmond Tutu Health Foundation, Sunnydale, Cape Town
  - JOSHA Research, Bloemfontein, Free State
  - Wits RHI, University of the Witwatersrand, Hillbrow, Johannesburg,Gauteng
  - Clinical HIV Research Unit (CHRU), Auckland Park, Johannesburg
  - Perinatal HIV Research Unit (PHRU), Diepkloof, Johannesburg
  - Setshaba Research Centre, Soshanguve, Tshwane
  - Groote Schuur Hospital, Cape Town, Western Cape
  - FAMCRU (Family Clinical Research with Ubuntu), Cape Town
  - Chatsworth, HIV Prevention Research Unit, South African Medical Research Council, Chatsworth
  - Isipingo, HIV Prevention Research Unit, South African Medical Research Council, Durban
  - Aurum Institute Tembisa, Tembisa
- University College London, London, United Kingdom
- Zambia (2):
  - Levy Mwanawasa University Teaching Hospital, Lusaka
  - Centre for Infectious Disease Research in Zambia [CIDRZ], Lusaka

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in the main publication may be shared, after de-identification.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: From 3 months after the last patient last visit onward.
Access Criteria: Investigators whose proposed use of the data has been approved by a review committee identified for this purpose.

REFERENCES:
- [Derived] Delany-Moretlwe S, Dehbi HM, Sikazwe I, Kyei G, Koram K, Dubberke E, Mwelase N, Hague D, Bekker LG, Yun L, Nel A, du Toit L, Biccard B, Gill K, Chipeta C, Mngadi KT, Lebina L, Dassaye R, Asari V, Fry SH, Turton E, Ahmed K, Kusi K, Adu-Amankwah S, Chilengi R, Chilekwa JC, Lovat L, McGuckin D, Caverly E, Politi M, Swan B, DeSchryver A, McKinnon S, Gupta A, Jones G, Freemantle N, Khader S, Rees H, Netea MG, Moonesinghe SR, Avidan MS. No evidence of MMR induced trained immunity to prevent SARS COV2: results from a multi-centre RCT. Front Immunol. 2025 Sep 16;16:1588190. doi: 10.3389/fimmu.2025.1588190. eCollection 2025. PMID 41035643
- [Derived] Noverr MC, Yano J, Hagensee ME, Lin HY, Meyaski MC, Meyaski E, Cameron J, Shellito J, Trauth A, Fidel PL Jr. Effect of MMR Vaccination to Mitigate Severe Sequelae Associated With COVID-19: Challenges and Lessons Learned. Med Res Arch. 2023 Feb;11(2):3598. doi: 10.18103/mra.v11i2.3598. PMID 37153751
- [Derived] Hirsch C, Park YS, Piechotta V, Chai KL, Estcourt LJ, Monsef I, Salomon S, Wood EM, So-Osman C, McQuilten Z, Spinner CD, Malin JJ, Stegemann M, Skoetz N, Kreuzberger N. SARS-CoV-2-neutralising monoclonal antibodies to prevent COVID-19. Cochrane Database Syst Rev. 2022 Jun 17;6(6):CD014945. doi: 10.1002/14651858.CD014945.pub2. PMID 35713300
- [Derived] Kreuzberger N, Hirsch C, Chai KL, Tomlinson E, Khosravi Z, Popp M, Neidhardt M, Piechotta V, Salomon S, Valk SJ, Monsef I, Schmaderer C, Wood EM, So-Osman C, Roberts DJ, McQuilten Z, Estcourt LJ, Skoetz N. SARS-CoV-2-neutralising monoclonal antibodies for treatment of COVID-19. Cochrane Database Syst Rev. 2021 Sep 2;9(9):CD013825. doi: 10.1002/14651858.CD013825.pub2. PMID 34473343

RESULTS

PARTICIPANT FLOW:
Groups:
- M-M-R II ®: Education and surveillance plus M-M-R II ®
  MR or M-M-R II ® vaccine: Education and surveillance plus MR or M-M-R II ® vaccine
- Placebo: Education and surveillance plus placebo
  Placebo: Placebo injection
Period: Overall Study
Arm/Group | M-M-R II ® | Placebo
Started (Number randomised) | 1722 | 1689
Completed (60 day follow-up for primary outcome) | 1607 | 1545
Not Completed | 115 | 144

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | M-M-R II ® | Placebo | Total
Number analyzed (Participants) | 1722 | 1689 | 3411
Age, Customized [Count of Participants; unit: Participants]
  <50 years | 1566 | 1539 | 3105
  >=50 years | 156 | 150 | 306
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1033 | 992 | 2025
  Male | 689 | 697 | 1386
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 85 | 68 | 153
  South Africa | 1252 | 1240 | 2492
  United Kingdom | 26 | 22 | 48
  Ghana | 76 | 75 | 151
  Zambia | 283 | 284 | 567

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Symptomatic COVID-19 at 60 Days
Description: Incidence of symptomatic (i.e. any of the following: cough, shortness of breath or difficulty breathing, fever, chills, muscle pain, sore throat, new loss of taste or smell, nausea, vomiting, or diarrhea), laboratory test-confirmed COVID-19 in the intervention and control groups in adults with repeated exposures to SARS-CoV-2 by day 60 after receiving trial intervention.
Time Frame: 60 days after receiving trial intervention
Measure: Count of Participants; unit: Participants
Arm/Group | M-M-R II ® | Placebo
Number analyzed (Participants) | 1607 | 1545
Participants | 24 | 19
Statistical Analysis 1: Comparison: M-M-R II ® vs Placebo; The primary endpoint was analysed using a Bayesian logistic regression, including as covariates the treatment arm, age (<50 vs. ≥50), and a random effect for site; Test type: Superiority; p = 0.52, Regression, Logistic; Risk Difference (RD) = 0.3, 95% CI 2-sided [-0.5 to 1.1]

2. Secondary Outcome: Number of Participants With Symptomatic COVID-19 at 150 Days
Description: Incidence of symptomatic (i.e. any of the following: cough, shortness of breath or difficulty breathing, fever, chills, muscle pain, sore throat, new loss of taste or smell, nausea, vomiting, or diarrhea), laboratory test-confirmed COVID-19 in the intervention and control groups in adults with repeated exposures to SARS-CoV-2 by day 150 after receiving trial intervention.
Time Frame: 150 days after receiving trial intervention
Measure: Count of Participants; unit: Participants
Arm/Group | M-M-R II ® | Placebo
Number analyzed (Participants) | 1585 | 1544
Participants | 65 | 64
Statistical Analysis 1: Comparison: M-M-R II ® vs Placebo; The endpoint was analysed using a Bayesian logistic regression, including as covariates the treatment arm, age (<50 vs. ≥50), and a random effect for site; Test type: Superiority; p = 0.95, Regression, Logistic; difference, 0·04%, 95% CI, -1·4% to 1·3%, p=0·95); Risk Difference (RD) = 0.04, 95% CI 2-sided [-1.4 to 1.3]

3. Secondary Outcome: Severity of COVID-19 Measured at 60 Days After Intervention
Description: Severity of COVID-19 in adults who become infected with SARS-CoV-2 by day 60 after receiving trial intervention. Severity will be graded on a simplified version of the ordinal WHO COVID-19 severity scale ((i) uninfected, (ii) infected but ambulatory [mild disease], (iii) infected and hospitalized [moderate or severe disease] or dead). Practically, this outcome measure was treated as a binary outcome - participants were classified and counted as having severe COVID-19 if they met the definition for the primary outcome of symptomatic COVID-19 AND were hospitalized during the course of their COVID-19 illness.
Time Frame: 60 days after receiving trial intervention
Measure: Count of Participants; unit: Participants
Arm/Group | M-M-R II ® | Placebo
Number analyzed (Participants) | 1607 | 1544
Participants | 3 | 1

4. Secondary Outcome: Severity of COVID-19 at 150 Days After Intervention
Description: Severity of COVID-19 in adults who become infected with SARS-CoV-2 by day 150 after receiving trial intervention. Severity will be graded on a simplified version of the ordinal WHO COVID-19 severity scale ((i) uninfected, (ii) infected but ambulatory [mild disease], (iii) infected and hospitalized [moderate or severe disease] or dead). Practically, this outcome measure was treated as a binary outcome - participants were classified and counted as having severe COVID-19 if they met the definition for the primary outcome of symptomatic COVID-19 AND were hospitalized during the course of their COVID-19 illness.
Time Frame: 150 days
Measure: Count of Participants; unit: Participants
Arm/Group | M-M-R II ® | Placebo
Number analyzed (Participants) | 1585 | 1544
Participants | 3 | 1

5. Secondary Outcome: Risk of SARS-CoV-2 Infection up to 150 Days After Trial Intervention
Description: Risk of SARS-CoV-2 infection by serology (anti-nucleocapsid antibody) in the intervention and control groups in adults with repeated exposures to SARS-CoV-2 by day 150 after receiving trial intervention. Infection with SARS CoV-2 during the course of the trial was diagnosed when IgG antibodies to the viral nucleocapsid protein were present from the 150 day specimen, but not the baseline specimen.
Time Frame: 150 days
Measure: Count of Participants; unit: Participants
Arm/Group | M-M-R II ® | Placebo
Number analyzed (Participants) | 945 | 951
Participants | 100 | 98

ADVERSE EVENTS:
Time Frame: 150 days from the date of administration of the investigational medicinal product
Description: Common Terminology Criteria for Adverse Events (CTACAE; v5.0 27-Nov-2017)
Arm/Group | M-M-R II ® | Placebo
All-Cause Mortality (participants affected / at risk) | 0/1722 | 0/1689
Serious Adverse Events (participants affected / at risk) | 11/1722 | 5/1689
Other Adverse Events (participants affected / at risk) | 0/1722 | 0/1689
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | M-M-R II ® (N=1722) | Placebo (N=1689)
COVID-19 (Infections and infestations) | 4 (4) | 1 (1)
Ovarian infection (Reproductive system and breast disorders) | 1 (2) | 0 (0)
Thromboembolic event (Cardiac disorders) | 1 (1) | 0 (0)
Suicide attempt (Psychiatric disorders) | 1 (1) | 0 (0)
Pre-eclampsia (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)
Right sided calcaneal fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 1 (1)
seizure (Nervous system disorders) | 0 (0) | 1 (1)
Pyrexia (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Tuberculous meningitis (Infections and infestations) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-10-12): https://cdn.clinicaltrials.gov/large-docs/32/NCT04333732/Prot_SAP_000.pdf
  • Informed Consent Form (2021-01-05): https://cdn.clinicaltrials.gov/large-docs/32/NCT04333732/ICF_001.pdf